CLINICAL TRIAL: NCT04066790
Title: A Randomised, Multicenter, Open-label, Phase II Study Evaluating Pyrotinib or Trastuzumab Plus Nab-paclitaxel as Neoadjuvant Therapy in Early Stage or Locally Advanced Human Epidermal Growth Factor Receptor (HER) 2 - Positive Breast Cancer
Brief Title: Pyrotinib or Trastuzumab Plus Nab-paclitaxel as Neoadjuvant Therapy in HER2-positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We terminated this trial and initiated a new one including pertuzumab.
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBC1901
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: HER2-positive; neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; 130-nm albumin-bound paclitaxel; Trastuzumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyrotinib in combination with nab-paclitaxel (Experimental): Prior to surgery: pyrotinib and nab-paclitaxel for 4 cycles (1 cycle = 21 days). After surgery/chemotherapy with epirubicin and cyclophosphamide (EC): trastuzumab up to 1 year total.
  Interventions: Drug: Pyrotinib; Drug: nab-Paclitaxel; Drug: Trastuzumab; Drug: EC chemotherapy; Procedure: Surgery
- Trastuzumab in combination with nab-paclitaxel (Active Comparator): Prior to surgery: trastuzumab and nab-paclitaxel for 4 cycles (1 cycle = 21 days). After surgery/chemotherapy with epirubicin and cyclophosphamide (EC): trastuzumab up to 1 year total.
  Interventions: Drug: nab-Paclitaxel; Drug: Trastuzumab; Drug: EC chemotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib 400 mg taken orally everyday, every 3 weeks, for 4 cycles.
  Arms: Pyrotinib in combination with nab-paclitaxel
Drug: nab-Paclitaxel — Nab-paclitaxel 100mg/m2 by intravenous (IV) infusion on day1, day8 and day15, every 3 weeks, for 4 cycles.
Drug: Trastuzumab — Trastuzumab IV infusion in 3-week cycles. Neoadjuvant treatment: 8 milligrams per kilogram (mg/kg) loading dose for Cycle 1, followed by 6 mg/kg for Cycles 2-4. Adjuvant treatment: 8 mg/kg loading dose for Cycle 9, followed by 6 mg/kg for remaining cycles till completion of 1 year trastuzumab
Drug: EC chemotherapy — epirubicin 90 mg/m2, and cyclophosphamide 600 mg/m2 by intravenous (IV) infusion every 3 weeks 4 cycles (Cycles 5-8)
Procedure: Surgery — All participants who are eligible for surgery will undergo surgery and have their pathologic response evaluated.

SUMMARY:
This study aims to evaluate the efficacy and safety of pyrotinib in combination with nab-paclitaxel or trastuzumab with nab-paclitaxel as neoadjuvant therapy in early stage or locally advanced HER2-positive breast cancer.

DETAILED DESCRIPTION:
The study evaluate the pathological complete response rate, event-free survival, disease-free survival, overall survival and safety of pyrotinib in combination with nab-paclitaxel or trastuzumab with nab-paclitaxel as neoadjuvant therapy in early stage or locally advanced HER2-positive breast cancer. Patients will receive 4 cycles of pyrotinib in combination with nab-paclitaxel or 4 cycles of trastuzumab with nab-paclitaxel as neoadjuvant therapy, then undergo surgery, then receive 4 cycles of epirubicin in combination with cyclophosphamide, then complete 1 year of trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* With signed consent
* Histologically confirmed invasive breast carcinoma with a primary tumor size of no less than (≥) 2 centimeters (cm) by standard local assessment technique
* Breast cancer stage at presentation: stage I-III
* HER2-positive breast cancer defined as 3+ score by immunohistochemistry in > 10 percent (%) of immunoreactive cells or HER2 gene amplification by in situ hybridization
* Known hormone receptor status (estrogen receptor and/or progesterone receptor)
* Eastern Cooperative Oncology Group Performance Status equal to or less than (<=) 1
* Baseline left ventricular ejection fracture >= 50% measured by echocardiography
* Willing to use highly effective form of nonhormonal contraception while on study and for 7 months after end of study treatment for female with fertility or male
* Negative serum pregnancy test for women with fertility
* Willing to obey the study protocol

Exclusion Criteria:

* Stage IV disease
* Previous anti-cancer therapy or radiotherapy for any malignancy
* History of other malignancy within 5 years prior to screening, except for appropriately-treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer
* Concurrent anti-cancer treatment in another investigational trial, including hormone therapy, bisphosphonate therapy, or immunotherapy
* Major surgical procedure unrelated to breast cancer within 4 weeks prior to randomization or from which the participant has not fully recovered
* Serious cardiac illness or medical condition
* Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness
* Any abnormalities in liver, kidney or hematologic function laboratory tests immediately prior to randomization
* Sensitivity to any of the study medications, any of the ingredients or excipients of these medications, or benzyl alcohol
* Not able to swallow the drug
* Pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Total Pathologic Complete Response (tpCR) | Cycle 4 . The duration of one treatment cycle is 21 days.
  tpCR is defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes after completion of neoadjuvant therapy and surgery (that is, ypT0/is, ypN0, in accordance with the current American Joint Committee on Cancer [AJCC] staging system).The duration of one treatment cycle is 21 days.

SECONDARY OUTCOMES:
Percentage of Participants With Breast Pathologic Complete Response (bpCR) | Cycle 4 . The duration of one treatment cycle is 21 days.
  bpCR is defined as the absence of any residual invasive cancer on the hematoxylin and eosin evaluation of the resected breast specimen after completion of neoadjuvant therapy and surgery (that is, ypT0/is, in accordance with current AJCC staging system).The duration of one treatment cycle is 21 days.
Clinical response | Cycle 4 . The duration of one treatment cycle is 21 days.
  Percentage of Participants With Complete Response, Partial Response, Stable Disease, or Progressive Disease During Cycles 1-4, According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. The duration of one treatment cycle is 21 days.
Event-free survival (EFS) | From Baseline to EFS event or date last known to be alive and event-free (up to 5 years)
  EFS is defined as the time from randomization to the first documentation of one of the following events: Disease progression (before surgery) as determined by the investigator with use of RECIST v1.1 Any evidence of contralateral disease in situ was not identified as progressive disease; Disease recurrence (local, regional, distant, or contralateral) after surgery; Death from any cause.
Disease-free survival (DFS) | From surgery to DFS event or date last known to be alive and event-free (up to 5 years)
  DFS was defined as the time from first date of no disease (i.e., date of surgery) to first documentation of one of the following events: Disease recurrence (local, regional, distant, or contralateral) after surgery. Any evidence of contralateral disease in situ was not identified as disease recurrence; Death from any cause.
Overall survival (OS) | From Baseline to OS event or date last known to be alive (up to 5 years)
  OS was defined as the time from randomization to death from any cause.

OTHER OUTCOMES:
Percentage of Participants With At Least One Adverse Event During Treatment Period | From randomization to 30 days after completion of study treatment
  The percentage of participants who experienced at least one adverse event during the neoadjuvant period, surgery, adjuvant treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No